CLINICAL TRIAL: NCT04155827
Title: Gender Specific Responses of Overweight and Obese Adults to Sprint Interval Training on Anthropometric Variables
Brief Title: Gender Specific Responses of Overweight and Obese Adults to Sprint Interval Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMFB1001
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIT for males (Experimental)
  Interventions: Other: SIT
- SIT for females (Experimental)
  Interventions: Other: SIT

INTERVENTIONS:
Other: SIT — Sprint interval training of 4*4, with 30 seconds of all out workout followed by 4 minutes of active recovery for 4 cycles.

SUMMARY:
Overweight and Obesity is a growing health problem worldwide. Lifestyle changes such as decreased physical activity, increased sedentary behaviour and unhealthy eating habits has contribute to this problem. According to World Health Organization (2016), more than 1.9 billion adults aged 18 years and older were overweight (39% of men and 40% of women).Regular exercise is the key contributor to energy expenditure and is essential for energy balance and weight control. Interval training (IT) has been commonly used for decades with purpose to improve body health and reduce weight loss and this exercise differs from the conventional aerobic exercise and endurance exercise as IT typically involves repeated bouts of relatively intense exercise interspersed by periods of lower- intensity effort or complete rest for recovery. One of the most common type of IT is sprint interval training (SIT). SIT involves 'supramaximal' effort (>100% VO2max) work bouts, traditionally structured as four to six 30s all-out effort and each round separated by 4 minutes of recovery period of a low intensity exercise. Potential physiological adaptation of SIT are highlighted by various studies reporting cardiovascular, skeletal muscle adaptations, increase fat oxidation that facilitate increases in both aerobic and anaerobic performance. In addition, SIT is able to improve maximal rate of oxygen consumption (VO2max), at the same time improving the peripheral vascular structure and function, enzymes of fat metabolism and increases insulin sensitivity. Previous SIT studies have included young healthy men and women, healthy obese young women, all of which have shown that SIT is effective for fat loss and improvement of some health parameters. However, whether SIT protocol is equally effective in improving the anthropometric measures in men and women remain unknown.

DETAILED DESCRIPTION:
Total of 80 eligible male (n=40) and female (n=40) young adults will be equally recruited using block randomization and chosen based on the inclusion and exclusion criteria. Before the study, all participants will be informed of the potential risks and benefits of the study. During the study period, participants will be instructed to avoid any form of physical activity besides the study protocol. Both groups will perform SIT protocol on a electromagnetically braked cycle ergometer three times per week for 6 weeks. Every session, participants start with a 5 minutes warm up at 50- 60% of heart rate maximum (HRmax) and follow by four 30-s all out bouts intersperse with 4 minutes of recovery (passive or no load cycling). For confirmation of all-out effort, participant are required to maintain his or her cycling cadence at least 60 rpm or above. Intervention will end with a 5 minutes cool down at 50- 60% of HRmax. Total duration for each session will be 28 minutes. If a participant misses fewer than three sessions per week non- consecutively, the sessions missed will be replace at the end of period. However, if participants misses three or more sessions, he or she will be excluded from the study. Outcome measures will be assessed at baseline and at end of 6 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI≧23kg/m2(WHO for Asia-Pacific region)
* No history of metabolic, hormonal, orthopedic, or cardiovascular diseases
* No current use of prescribed medication including oral contraception

Exclusion Criteria:

* Contraindications to physical activity assessed by Physical Activity Readiness Questionnaire-PAR-Q
* Undergoes any surgical or hormone treatment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Both genders (male & female) will be equally recruited.
Enrollment: 35 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
BMI for change | At baseline (before intervention begin) and post training (end of 6 weeks).
Waist Circumference for change | At baseline (before intervention begin) and post training (end of 6 weeks).
Total Fat % for change | At baseline (before intervention begin) and post training (end of 6 weeks).
Lean Muscle Mass for change | At baseline (before intervention begin) and post training (end of 6 weeks).
skin Fold Measurement for change | At baseline (before intervention begin) and post training (end of 6 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Imtiyaz Ali Mir, Principal Investigator — Universiti Tunku Abdul Rahman
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No